CLINICAL TRIAL: NCT02159911
Title: Use of Oral Misoprostol for Cervical Priming Before Hysteroscopy: a Randomized Comparison of Two Dosages
Brief Title: Oral Misoprostol for Cervical Priming Before Hysteroscopy
Status: Completed | Type: Observational
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Other Study IDs: USJ-002
Record Dates: First submitted 2014-06-02; First posted 2014-06-10 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Cervical Laceration; Adverse Effects
Keywords: Cervical; Hysteroscopy; Misoprostol; Oral
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 200 mcg misoprostol: Misoprostol administered orally one hour before surgery
  Interventions: Drug: Misoprostol administered orally one hour before surgery
- 400 mcg misoprostol: Misoprostol administered orally one hour before surgery
  Interventions: Drug: Misoprostol administered orally one hour before surgery

INTERVENTIONS:
Drug: Misoprostol administered orally one hour before surgery — Closed and numbered envelopes, containing a capsule with either 200mcg or 400mcg of misoprostol were randomly distributed to the patients. Each envelope was coded randomly and only the pharmaceutical department of the hospital knew the content of these envelopes and kept a list of their codes.
  The misoprostol was administered by the floor nurse, per-os to the patient one hour before hysteroscopy with a small amount of water. The number on the envelope was noted by the nurse on the document relative to the patient. Hence, the patient, the physician performing the biopsy, the nurse and the research associate did not know the exact dose of misoprostol that was ingested by the patient.
  Other Names: ( Cytotec*)

SUMMARY:
A randomized, double blind study to compare 200 and 400 mcg misoprostol for cervical preparation before hysteroscopy.

DETAILED DESCRIPTION:
All patients admitted for hysteroscopy were offered participation in the study, and those choosing to participate were assessed according to the inclusion and exclusion criteria of the study protocol. The investigators included all non pregnant patients who were considered medically fit and scheduled for operative hysteroscopy, regardless of age or indication of the hysteroscopy. Patients with a positive history of vascular or coronary artery disease and patients using other products that could affect the consistency of the cervix such as local estrogen or laminaire were excluded from the study. To achieve a mean difference of 0.5 in the diffculty of dilation and a mean difference of 0.5 in the First Hegar with a power of 80% at 0.05 statistical significance, a sample of 163 patients in each arm is needed. However, the investigators patients pool did not permit to recruit more than 70 women so the investigators took it as a convenience sample of a total of 70 women that agreed to be recruited for the trial. An informed consent was obtained after explaining to the patients the benefit and the eventual risk or adverse effects associated with the medication. Studied factors were: age, parity, reason for the procedure, history of cervical dilation and history of cervical surgery.

Seventy closed and numbered envelopes, containing a capsule with either 200mcg or 400mcg of misoprostol were randomly distributed to these 70 patients. Each envelope was coded randomly and only the pharmaceutical department of the hospital knew the content of these envelopes and kept a list of their codes.

The misoprostol was administered by the floor nurse, per-os to the patient one hour before hysteroscopy with a small amount of water. The number on the envelope was noted by the nurse on the document relative to the patient. Hence, the patient, the physician performing the biopsy, the nurse and the research associate did not know the exact dose of misoprostol that was ingested by the patient.

Three physicians contributed to the study. Before beginning the procedure, the operator noted by pelvic examination the position of the cervix. He then noted the size/number of the first Hegar dilator used, the maximal dilation reached, the difficulty to dilate during the intervention (measured by a scale from 1 to 10), cervical injuries, bleeding or uterine perforation and the duration of the operation. A rigid hysteroscope (Storz, 27 F) was used for all procedures.

Adverse effects that could be related to misoprostol (uterine cramps, nausea, vomiting, diarrhea and fever), were reported before and up to 6 hours after surgery.

Statistical analysis was performed using SPSS version 18. Means comparison was done using t-test for continuous variables such as difficulty in dilation or first Hegar (the data was normally distributed). Frequency and percent distribution were compared between the two treatment groups using χ2 test when the expected cell count was 5 or more; in cases where the expected cell count was less than 5, the Fisher exact test was used instead

ELIGIBILITY:
Inclusion Criteria:

* non pregnant patients
* considered medically fit without any life threatening conditions
* scheduled for operative hysteroscopy, regardless of age or indication of the hysteroscopy

Exclusion Criteria:

* a positive history of vascular or coronary artery disease
* using other products that could affect the consistency of the cervix such as local estrogen or laminaire

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted for hysteroscopy were offered participation in the study, and those choosing to participate were assessed according to the inclusion and exclusion criteria of the study protocol
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2004-06; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Ease of cervical dilatation | Assessed during the surgery and recorded immediately at the end of surgery
  Measured by a scale from 1 to 10

SECONDARY OUTCOMES:
Adverse effects | recorded till 6 h following surgery
  uterine cramps, nausea, vomiting, diarrhea and fever

OTHER OUTCOMES:
Complications during hysteroscopy | recorded immediately at the end of surgery
  cervical injuries, bleeding or uterine perforation

CONTACTS AND LOCATIONS:
Overall Officials: Assaad K Kesrouani, MD, Principal Investigator — Saint-Joseph University
Locations (1):
- Hotel-Dieu de France University Hospital, Beirut, Lebanon, Lebanon

REFERENCES:
- [Result] Lee YY, Kim TJ, Kang H, Choi CH, Lee JW, Kim BG, Bae DS. The use of misoprostol before hysteroscopic surgery in non-pregnant premenopausal women: a randomized comparison of sublingual, oral and vaginal administrations. Hum Reprod. 2010 Aug;25(8):1942-8. doi: 10.1093/humrep/deq083. Epub 2010 Jun 11. PMID 20542898
- [Result] Bastu E, Celik C, Nehir A, Dogan M, Yuksel B, Ergun B. Cervical priming before diagnostic operative hysteroscopy in infertile women: a randomized, double-blind, controlled comparison of 2 vaginal misoprostol doses. Int Surg. 2013 Apr-Jun;98(2):140-4. doi: 10.9738/INTSURG-D-12-00024.1. PMID 23701149